CLINICAL TRIAL: NCT00685906
Title: A Randomised, Double-blind, Two-way Crossover Study to Determine the Effects of Co-administration of AZD6140 and Nordette® (Combination of Levonorgestrel and Ethinyl Estradiol) After Multiple Oral Doses in Healthy Female Volunteers
Brief Title: AZD6140 Oral Contraceptive Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jay Horrow, MD, Medical Science Director, AZD6140, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D5130C00042; AZD6140/OC Study
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: oral contraceptive; birth control; Healthy volunteers
MeSH Terms: interventions — Ticagrelor; Levonorgestrel; Ethinyl Estradiol; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD6140
- 2 (Active Comparator)
  Interventions: Drug: Levonorgestrel and Ethinyl Estradiol (Nordette®)

INTERVENTIONS:
Drug: AZD6140 — 90 mg tablet taken by mouth 2 times a day for 21 days per cycle
  Arms: 1
Drug: Levonorgestrel and Ethinyl Estradiol (Nordette®) — 1 tablet taken by mouth once a day for 28 days per cycle
  Other Names: Nordette®
  Arms: 2

SUMMARY:
The purpose of this study is to examine the effect of co-administration of AZD6140 and Nordette® on the blood levels of certain female hormones.

ELIGIBILITY:
Inclusion Criteria:

* Females who are healthy, non-pregnant, not planning pregnancy within the study period, non-breast-feeding, and pre-menopausal
* Either currently taking Nordette® which was well tolerated for at least two months prior to randomisation with no history of break-through bleeding, or, willing to take Nordette for 2 months prior to receiving the study drug
* Females of child-bearing potential must be willing to use at least 1 additional medically approved non-hormonal barrier contraceptive method (for example, condom or diaphragm) that contains spermicide

Exclusion Criteria:

* History of intolerance (e.g. adverse events) to any oral contraceptive or AZD6140
* History of blood vessel or bleeding conditions that would make the volunteer more prone to bleeding
* History or presence of significant medical problems
* Women who are current smokers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Blood levels of ethinyl estradiol, a female hormone, following oral administration of AZD6140 and Nordette® | At scheduled times following dosing during the first 3 weeks of menstrual cycles 1 and 2.

SECONDARY OUTCOMES:
Blood levels of various other hormones following concomitant oral administration of AZD6140 and Nordette® | At scheduled times following dosing during the first 3 weeks of menstrual cycles 1 and 2.
Blood levels of AZD6140 and its main metabolite after concomitant oral administration of AZD6140 and Nordette® | At scheduled times following dosing during the first 3 weeks of Cycles 1 and 2.
Safety and tolerability of AZD6140 when co-administered with Nordette® | Screening through completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — AstraZeneca; Audrey, Martinez, MD, Principal Investigator — SeaView Research
Locations (1):
- Research Site, Miami, Florida, United States